CLINICAL TRIAL: NCT00006552
Title: Adherence to Antihypertensive Therapy--Data Analyses
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 953; R03HL064273 (NIH)
Record Dates: First submitted 2000-11-28; First posted 2000-11-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To assess factors that may influence adherence to antihypertensive drug therapy.

DETAILED DESCRIPTION:
BACKGROUND:

High blood pressure continues to be a highly prevalent condition affecting about 20 percent of the U.S. population. Untreated, it may lead to coronary heart disease, stroke, kidney failure, and other complications. Medication is a major means of controlling hypertension and averting these debilitating consequences. Treatment with drugs, however, is undermined by suboptimal adherence to therapy. Forgetting to take medications is the most commonly elicited reason for lapses in medication use; but side effects, health beliefs, lack of knowledge of disease and treatment instructions, and financial barriers may also interfere. Determining those factors that (1) are predictably associated with fluctuations in adherence (such as day of the week, holidays, medication appointments); (2) ameliorate the impact of nonadherence, such as pharmacologic properties of drugs that protect patients during adherence lapses; and (3) correlate with the accuracy of adherence reporting by patients will assist in anticipating and addressing adherence obstacles and serve as the objectives of the study.

DESIGN NARRATIVE:

The study used data collected from electronic adherence monitors, questionnaires, and computerized medical records that contained blood pressure readings during a prior investigation of antihypertensive adherence. This earlier investigation, conducted from 1994 to 1997, involved 286 members of Harvard Pilgrim Health Care who were on single drug therapy for mild to moderate hypertension. Objective 1 evaluated the impact of temporal factors such as weekend versus weekday, holidays, seasons, and impending medical appointments on adherence by analyzing their effects on the daily rate of dosing recorded by electronic medication monitors. Time trend models were used for this purpose. Objective 2 assessed the impact of pharmacologic duration of action on the level of antihypertensive adherence required to maintain a goal blood pressure of <140/90 mmHg. This involved determining if the relationship between adherence and blood pressure was modified by the duration of drug effect. Objective 3 concerning correlates of accuracy of reported adherence was approached by verifying reported adherence against electronically measured adherence. Predictors and correlates of accurately reported adherence such as patient age, gender, race/ethnicity, education, socioeconomic status, health beliefs, and measures of health status were then identified by cross tabulating and statistical modeling accurate reporting against these factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Choo — Brigham and Women's Hospital

REFERENCES:
- [Background] Choo PW, Rand CS, Inui TS, Lee ML, Canning C, Platt R. A cohort study of possible risk factors for over-reporting of antihypertensive adherence. BMC Cardiovasc Disord. 2001;1:6. doi: 10.1186/1471-2261-1-6. Epub 2001 Dec 13. PMID 11801191
- [Background] Choo PW, Rand CS, Inui TS, Lee ML, Ma CC, Platt R. A pharmacodynamic assessment of the impact of antihypertensive non-adherence on blood pressure control. Pharmacoepidemiol Drug Saf. 2000 Dec;9(7):557-63. doi: 10.1002/pds.539. PMID 11338913